CLINICAL TRIAL: NCT04556292
Title: A Phase 2, Open-Label, Multi-Center Study of SC10914 in Germline BRCA Mutation Subjects With Locally Advanced and/or Metastatic Breast Cancer, Who Have Received More Than 2 Prior Chemotherapy Regimens for Metastatic Disease
Brief Title: A Phase II Study to Assess the Efficacy and Safety of SC10914 in the Metastatic Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QF-SC10914-203
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer Metastatic; BRCA 1 Gene Mutation; BRCA 2 Gene Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SC10914 group (Experimental)
  Interventions: Drug: SC10914

INTERVENTIONS:
Drug: SC10914 — SC10914 400mg tid

SUMMARY:
This open label, multi-centre phase II study will assess the efficacy and safety of single agent SC10914 in metastatic breast cancer patients with gBRCA 1/2 mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Germline mutation in BRCA1 or BRCA2
2. Histologically or cytologically confirmed breast cancer with evidence of metastatic disease.
3. Prior therapy with an anthracycline and/or a taxane in either an adjuvant or metastatic setting
4. Patients who have received platinum (cisplatin or carboplatin, either as monotherapy or in combination) for advanced breast cancer are eligible to enter the study provided platinum-free interval at least 6 months (time from last dose of platinum chemotherapy to disease progression
5. Patients who have received platinum as potentially curative treatment for a prior cancer (e.g. ovarian cancer) or as adjuvant/neoadjuvant treatment for breast cancer are eligible provided at least 12 months have elapsed between the last dose of platinum-based treatment and eligible .
6. Patients with estrogen and/or progesterone receptor-positive disease must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy .
7. At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT (MRI where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1.
8. ECOG performance status 0-1.
9. Adequate bone marrow, kidney and liver function

Exclusion Criteria:

1. Prior treatment with PARP inhibitor.
2. Patients with HER2 positive disease
3. Untreated and/or uncontrolled brain metastases
4. Known HIV (Human Immunodeficiency Virus) infection.
5. Persistent toxicities (≥CTCAE grade 2) caused by previous cancer therapy, excluding alopecia
6. Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to a maximum of 30 months
  Using Independent Central Review Data Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Assessed up to a maximum of 30 months
  Using Independent Central Review According to Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1)
Overall Survival (OS) | Assessed up to a maximum of 30 months
  from eligible until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: hu xichun, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No